CLINICAL TRIAL: NCT03320421
Title: Phase II Trial of Hypofractionated Whole-breast Radiation and Concomitant Boost to the Surgical Bed After Breast Conserving Surgery
Brief Title: Hypofractionated Radiation Therapy With Concomitant Boost in Treating Women After Breast Conserving Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Yu Tang, Doctor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2016YQ-19
Record Dates: First submitted 2017-07-25; First posted 2017-10-25 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer Female
Keywords: hypofractionated radiation; breast cancer; breast conserving surgery; simultaneous boost radiation
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIB group (Experimental): Radiation therapy:
  daily 5 days per week for 3 weeks. 43.5 Gy in 15 fractions to the whole breast 49.5 Gy in 15 fractions to the tumor bed boost
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Radiation to the whole breast: 43.5 Gy in 15 fractions in 3 weeks. Simultaneous radiation to the surgical cavity: 49.5 Gy in 15 fractions in 3 weeks.
  Intensity modulated radiation treatment is used.

SUMMARY:
This phase II study is to evaluate the safety of hypofractionated whole breast radiation (HFRT) with simultaneous tumor bed boost(SIB) in women with early breast cancer after breast-conserving surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

To determine the toxicity with adjuvant hypofractionated whole breast radiation with simultaneous tumor bed boost (SIB) in women with early breast cancer after breast conserving surgery.

Secondary:

To determine the short term cosmetic and quality of life of the participants treated with this regimen.

To determine the local control of the participants treated with this regimen.

OUTLINE: Patients undergo adjuvant hypofractionated whole breast radiation with simultaneous tumor bed boost once daily a week for 3 weeks. Toxicity, quality of life and cosmetic result is assessed before radiation, at the end of the radiation, within 2, 4, 6 weeks after completion of radiotherapy, and then every 3 months for 1 ear.

PROJECTED ACCRUAL: A total of 90 participants will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* female, aged between 18-70
* pathological confirmed breast invasive carcinoma
* patients after breast lumpectomy(including quadrantectomy) with axillary lymph nodes dissection or sentinel node biopsy
* stage p T 1-2 N 0
* metastasis omitted by routine examinations in 1 months before enrollment
* complete blood count obtained in 2 weeks prior to study entry should meet the following criteria: absolute neutrophil count > 1.8 *10^9/L, hemoglobin > 8.0g/dl, platelet > 75 * 10^9/L
* hepatic and renal function in 2 weeks prior to study entry should be normal
* study entry within 60 days from whichever comes later: surgery or last chemotherapy
* women of childbearing potential must have a negative urine or serum pregnancy test with 2 weeks of study entry
* signs study specific informed consent prior to study entry

Exclusion Criteria:

* breast cancer with stage III/III (AJCC 7th)
* occult breast cancer
* in-situ breast carcinoma
* bilateral breast cancer
* male breast cancer
* breast lymphoma or breast sarcoma
* combined with Paget's disease
* received preoperative treatment(including neoadjuvant chemotherapy, endocrine therapy and target therapy
* positive surgical margin
* axillary lymph nodes dissection or sentinel lymph node biopsy omitted
* regional lymph nodes radiation needed
* boost volume larger than 1/4 of the whole breast
* tumor bed unable to recognize on CT
* prior invasive malignant tumor history
* prior radiation to thoracic
* connective tissue disease, such as active systemic lupus erythematosus and scleroderma, etc.
* severe, active co-morbidity, defined as follows:

  * unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * severe, acute bacterial or fungal infection within the last 2 weeks
  * chronic obstructive pulmonary disease exacerbation or other respiratory illness within 30 days
* pregnant women

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
acute radiation induced dermatitis by CTCAE within 3 months | 3 months
  radiation induced skin toxicity, including rash, dry skin, ulceration etc., occurring immediately after radiation.

SECONDARY OUTCOMES:
late radiation toxicity by CTCAE every 3 months to 1 years after 3 months of completion of radiation | 3 months to 1 year
  any radiation induced toxicity occurring after the radiation
breast cosmetic result as measured by Harvard scale of breast cosmesis (excellent, good, fair, poor) every 3 months for 1year | every 3 months for 1year
  breast cosmetic evaluation after breast conserving surgery and radiation, using Harvard scale.
quality of life as measured by Functional Assessment of Cancer Therapy-Breast Scale (FACT-B) every 3 months for 1 year | every 3 months for 1 year
  Functional Assessment of Cancer Therapy-Breast Scale (FACT-B) is used to evaluated the quality of life: all scale range: 0-144; sub-scale range: physical well being: 0-28; social well being: 0-28; emotional well being 0-24; functional well being 0-28; additional consideration: 0-36; the higher the better
quality of life as measured by Breast Cancer Treatment Outcome Scale(BCTOS) every 3 months for 1 year | every 3 months for 1 year
  Functional Assessment of Breast Cancer Treatment Outcome Scale(BCTOS) is used to evaluated the quality of life. the range of BCTOS is 22-88, the smaller the better
in-breast recurrence rate at 1 year of radiation completion | 1 year
  recurrence occurred in the treated breast.

CONTACTS AND LOCATIONS:
Overall Officials: Yexiong Li, Professor, Principal Investigator — Cancer Hospital/Institution, Chinese Academic Medical Sciences and Peking Union Medical College
Locations (1):
- National Cancer Center/Cancer Hosptial, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Darby S, McGale P, Correa C, Taylor C, Arriagada R, Clarke M, Cutter D, Davies C, Ewertz M, Godwin J, Gray R, Pierce L, Whelan T, Wang Y, Peto R. Effect of radiotherapy after breast-conserving surgery on 10-year recurrence and 15-year breast cancer death: meta-analysis of individual patient data for 10,801 women in 17 randomised trials. Lancet. 2011 Nov 12;378(9804):1707-16. doi: 10.1016/S0140-6736(11)61629-2. Epub 2011 Oct 19. PMID 22019144
- [Background] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial A of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet Oncol. 2008 Apr;9(4):331-41. doi: 10.1016/S1470-2045(08)70077-9. Epub 2008 Mar 19. PMID 18356109
- [Background] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bentzen SM, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial B of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet. 2008 Mar 29;371(9618):1098-107. doi: 10.1016/S0140-6736(08)60348-7. Epub 2008 Mar 19. PMID 18355913
- [Background] Whelan TJ, Pignol JP, Levine MN, Julian JA, MacKenzie R, Parpia S, Shelley W, Grimard L, Bowen J, Lukka H, Perera F, Fyles A, Schneider K, Gulavita S, Freeman C. Long-term results of hypofractionated radiation therapy for breast cancer. N Engl J Med. 2010 Feb 11;362(6):513-20. doi: 10.1056/NEJMoa0906260. PMID 20147717
- [Background] Hamilton DG, Bale R, Jones C, Fitzgerald E, Khor R, Knight K, Wasiak J. Impact of tumour bed boost integration on acute and late toxicity in patients with breast cancer: A systematic review. Breast. 2016 Jun;27:126-35. doi: 10.1016/j.breast.2016.03.002. Epub 2016 Apr 22. PMID 27113229
- [Background] Chadha M, Vongtama D, Friedmann P, Parris C, Boolbol SK, Woode R, Harrison LB. Comparative acute toxicity from whole breast irradiation using 3-week accelerated schedule with concomitant boost and the 6.5-week conventional schedule with sequential boost for early-stage breast cancer. Clin Breast Cancer. 2012 Feb;12(1):57-62. doi: 10.1016/j.clbc.2011.09.002. Epub 2011 Nov 6. PMID 22056970
- [Background] Cante D, Franco P, Sciacero P, Girelli G, Marra AM, Pasquino M, Russo G, Borca VC, Mondini G, Paino O, Barmasse R, Tofani S, Numico G, La Porta MR, Ricardi U. Five-year results of a prospective case series of accelerated hypofractionated whole breast radiation with concomitant boost to the surgical bed after conserving surgery for early breast cancer. Med Oncol. 2013 Jun;30(2):518. doi: 10.1007/s12032-013-0518-7. Epub 2013 Mar 5. PMID 23460537
- [Background] Freedman GM, White JR, Arthur DW, Allen Li X, Vicini FA. Accelerated fractionation with a concurrent boost for early stage breast cancer. Radiother Oncol. 2013 Jan;106(1):15-20. doi: 10.1016/j.radonc.2012.12.001. Epub 2013 Jan 17. PMID 23333014